CLINICAL TRIAL: NCT06704633
Title: Health Status After Switching Angiotensin-converting Enzyme Inhibitors or Angiotensin Receptor Blockers to Sacubitril-valsartan in Patients With Heart Failure With Reduced Ejection Fraction From Rural Tanzania: An Interventional Study
Brief Title: Sacubitril-valsartan in Patients With Heart Failure With Reduced Ejection Fraction From Rural Tanzania
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Martin Rohacek (Other)
Collaborators: Ifakara Health Institute (IHI) (Unknown)
Responsible Party: Sponsor-Investigator, Martin Rohacek, Project Leader, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-50 Heart failure Tz
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
Keywords: Sacubitril-valsartan; Heart failure with reduced ejection fraction,; HFrEF; KCCQ
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: This is an interventional single center single group open label pre-post study with a follow-up of 10 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Symptomatic adult particiopants with HFrEF, under heart failure therapy (Other): Symptomatic adults with HFrEF, under heart failure medication
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet — A 36-hour wash-out of ACE inhibitors before initiating ARNI will be done, because of a risk of angioedema if ARNI is started without a wash-out period. The ACE inhibitor or ARB will be switched to sacubitril/valsartan 50mg twice daily (24.3 mg sacubitril, 25.7mg valsartan) for two weeks, increased to 100mg twice daily for three weeks, followed by 200mg twice daily

SUMMARY:
Angiotensin-neprilysin inhibitors (ARNI) are beneficial in patients with heart failure with reduced ejection fraction. No study evaluating ARNI has been conducted in sub-Saharan Africa (except South Africa) yet, where heart failure is a major health problem. Before implementing ARNI in Tanzania, a study evaluating the benefit and safety of ARNI in Africans is needed. The aim of this interventional pre-post study is to evaluate the health status of symptomatic patients with heart failure with reduced ejection fraction who are under a chronic heart failure therapy, before and after switching angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARB) to ARNI. Participants will be recruited at the Heart and Lung Clinic of the St Francis Regional Referral Hospital in Ifakara in rural Tanzania during a study period of 30 months, including 10 months of follow-up. A total of 238 participants will be included. The investigators hypothesize that health status, expressed by the Kansas City Cardiomyopathy Questionnaire summary score and 6-minute walking test, will improve after switching from ACE-inhibitors or ARB to ARNI. In Tanzania, sacubitril/valsartan is registered under the name Uperio®.

DETAILED DESCRIPTION:
Background Non-communicable diseases (NCDs) cause more than 40 million deaths globally each year, and more than three quarters of them occur in low- and middle-income countries. The majority of deaths are caused by cardiovascular diseases, such as heart failure and stroke. Mortality from heart failure has been reported to be highest in Africa, with a one-year mortality rate of 34% compared to 16.5% in other low- and middle-income countries. Arterial hypertension is the most common underlying risk factor for heart failure in sub-Saharan Africa, also in rural areas. Patients mostly present in advanced stages of heart failure, and are not under regular treatment. International guidelines recommend diuretics, angiotensin- converting enzyme (ACE) inhibitors or angiotensin-neprilysin inhibitors (ARNI), angiotensin 2 receptor blockers (ARB), if ACE-inhibitors are not tolerated, beta-blockers, mineralocorticoid receptor antagonists, and sodium glucose co- transporter 2 (SGLT-2) inhibitors for treatment of chronic heart failure with reduced ejection fraction. An intensive treatment strategy with rapid up-titration of guideline-directed chronic heart failure therapy after acute heart failure reduces symptoms, improves quality of life, reduces the risk for all cause death, and is well tolerated. The PARADIGM trial showed that, if enalapril 10mg twice daily for at least 2 weeks was switched to sacubitril/valsartan in symptomatic patients with a left ventricular ejection fraction (LVEF) of ≤40% who had been under a stable heart failure therapy for at least 4 weeks, the combined endpoint of death and hospitalization for heart failure was significantly reduced from 26.5% to 21.8% compared to if the ACE inhibitor was continued. In the CHAMP-HF, a multicenter observational study of American outpatients with heart failure with reduced ejection fraction (HFrEF), 35.8% patients initiated on ARNI had a large (10 to <20 points) or very large (20 points and more out of 100) improvement in their health status expressed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) summary score measured by the KCCQ-12 short version over a median (IQR) of 10.7 (6.7 -11.7) months of follow up, vs 27.5% of patients not initiated on ARNI. Among patients with HFrEF who were hospitalized for acute decompensated heart failure, the initiation of sacubitril/valsartan therapy led to a greater reduction in the N-terminal pro brain natriuretic peptide (NT-proBNP) blood concentration than enalapril therapy. One study could not detect any racial and ethnic differences in reduction of NT-proBNP, improvement in health status, and reverse remodeling in patients with systolic heart failure treated with sacubitril/valsartan. In patients with salt-sensitive hypertension, sacubitril/valsartan was superior to valsartan in office- and ambulatory blood pressure control, and was associated with an increased natriuresis and diuresis. Moreover, sacubitril-valsartan had a positive effect on glycemic control of heart failure patients with diabetes mellitus. It had similar effect on kidney function and albuminuria in patients with chronic renal failure compared to irbesartan.

In the PARADIGM trial, participants were recruited also in South Africa. However, none of the other studies were done in Africa, and the efficacy and safety of sacubitril/valsartan has never been studied in African patients outside South Africa. Sacubitril/valsartan is registered in Tanzania under the product name Uperio®.

The investigators hypothesize that the switch from a well-dosed ACE inhibitor or ARB to sacubitril/valsartan leads to an improvement of the health status, to an increase in the 6-minute walking distance, and to a reduction of the brain natriuretic peptide (BNP) blood concentration, in symptomatic patients with heart failure with reduced ejection fraction (HFrEF) from sub-Saharan Africa who are under a stable chronic heart failure therapy.

Setting The study will be conducted at the St Francis Regional Referral Hospital, Ifakara. This hospital is a referral center for a population of about 1 million people living in the Kilombero valley in rural Tanzania. Since 2021, a Heart and Lung Clinic has been annually serving 5000 patients with heart - or lung diseases. Comprehensive echocardiography, electrocardiography, lung ultrasound, and laboratory tests are done on a routine basis by a trained team. A patients cohort including more than 800 patients has been established. Sacubitril/valsartan is not prescribed yet for patients attending the clinic. The laboratory of the hospital offers chemistry including the measurement of serum-BNP routinely. There is an oxygen plant, an emergency department managing 90'000 patients per year, and a high dependency unit caring for 500 patients per year in this hospital.

Sample size Sample size calculation is based on a study which reported that 35.8% of patients receiving ARNI experienced a large (≥10-points) or very large (≥20-points) improvement in the KCCQ summary score, compared to 27.5% of patients not initiated on ARNI therapy. Based on these effect sizes, the investigators calculated that a sample size of 238 patients would be required to detect a statistically significant difference with 80% power and a two-sided test at a 5% significance level, accounting for an expected 25% rate of mortality or loss to follow-up.

Study procedures Patients will be screened in the Heart and Lung Clinic of the St Francis Regional Referral Hospital, and participants already included in the patient cohort of the Heart and Lung Clinic will be contacted and invited to participate. Before enrolment, the heart failure medication of potentially eligible patients will be optimized (i.e diuretics adapted to volume status, ACE inhibitors or ARB, betablockers, and spironolactone increased to high therapeutic doses (lisinopril to at least 10mg once daily or enalapril at least 10mg twice per day, losartan at least 50mg once daily, carvedilol at least 12.5mg twice per day or bisoprolol at least 5mg once daily, and spironolactone at least 25mg once daily). Adherence will be assessed by pill count and self-report.

Newly diagnosed untreated patients with heart failure will be started on heart failure therapy, rapidly up titrated, and invited to be reevaluated for enrolment after 3 months. At enrolment, patients will sign an informed consent, and will be instructed to continue to adhere to prescribed therapy. The following baseline examinations will be done: history taking including adherence to medication, physical examination including standardized blood pressure measurement, and oxygen saturation, KCCQ summary score measured by the KCCQ-12 version which was validated in Tanzania, comprehensive echocardiography, electrocardiography, and 6-minute walking test will be done according to standard operating procedures. Blood samples for hemoglobin, random glucose, brain natriuretic peptide (BNP), creatinine, liver enzymes, HIV, and electrolytes (potassium, sodium, calcium) will be taken. A 36-hour wash-out of ACE inhibitors before initiating sacubitril/valsartan will be done, because of a risk of angioedema if sacubitril/valsartan is started without a wash-out period. The ACE inhibitor or ARB will be switched to sacubitril/valsartan 50mg twice daily (24.3 mg sacubitril, 25.7mg valsartan) for two weeks, increased to 100mg twice daily for three weeks, followed by 200mg twice daily. Betablocker and spironolactone will be continued, and diuretics dosages adapted as clinically indicated. Follow-up visits will be done after 2 weeks, 5 weeks, 2 months, 4 months, 6 months and 10 months after switching to sacubitril/valsartan including history taking and physical examination. Adherence to medication will be assessed by pill count and self-report. KCCQ summary score and 6-minute walking test will be done after 5 weeks, 2-, 4-, 6-, and 10 months, creatinine and electrolytes will be measured in serum after 5 weeks, and after 4-, and 10 months, and BNP after 10 months of follow-up.

Echocardiography will be performed at 6 months and 10 months follow-up visits. The echocardiographer doing follow-up echocardiography will be blinded to the result of the baseline echocardiogram.

The cost for the routine guideline directed heart failure medication (diuretics, ACE-inhibitors, ARB, betablocker, spironolactone) will be covered by health insurance or by the participant. Sacubitril-valsartan will be provided by Novartis. Transport costs for the follow-up visits will be reimbursed. After the end of the study, sacubitril/valsartan will be available for the patients for a price comparable to locally available ACE-inhibitors.

Statistical analysis Descriptive statistical analysis will be used to describe primary and secondary outcomes. The proportion of participants with a large (≥10 points) or very large (≥20 points) improvement in KCCQ summary score from baseline to after 5 weeks, 2, 4, 6, and 10 months of follow-up will be calculated. Plots displaying the adjusted estimated mean KCCQ score and confidence limits over time from restricted cubic splines regression will be presented. The median changes in KCCQ summary score, NYHA class, distance in the 6-minute walking test, BNP and left ventricular ejection fraction (LVEF) from baseline to after 5 weeks, 2, 4, 6, and 10 months of follow-up will be calculated. Time to death or lost to follow up will be estimated using Kaplan-Meier methods. All estimates will be reported using 95% confidence intervals and a p-value ≤0.05 will be considered statistically significant.

Data Management All data will be managed using the same data collecting system (RedCap). Data will stored using the RedCap server of the Ifakara Health Institute, using a computer with double password protection. Data extraction is done daily and stored on a secured cloud storage service (IHI-drive, and on switchdrive for back-up (https://drive.switch.ch) accessible only by study team members through a username-password authentication. Thus, data can be handled securely during the project. All folder structures and naming conventions will be generated by the responsible investigators, and all project members will be instructed in how to fill in the data by the responsible investigators.

Data security Security standard will be adopted from the ISO 27001-Information security management. All participants data will be coded, and all data will be password secured. Thus, the data security will be high. All study related data will be stored in the IHI server as per institution protocol.

Ethical Clearance The protocol will be submitted to the Ethikkomission der Nord-und Zentralschweiz, Switzerland, the institutional Review Board of the Ifakara Health Institute, and the Ethical Committee of the National Institute for Medical Research, Tanzania (NIMR), and Tanzania Commission for Science and Technology (COSTECH). Patients will be only be included, if they agree and after having signed written informed consent.

Risks Sacubitril/Vasartan has been studied in large randomized controlled trials, and been approved by food and drug administrations and registered worldwide. In Tanzania, sacubitril/valsartan is prescribed, and registered under the name Uperio®. We do not expect more side effects than have been described already in previous trials. Since about 5000 patients are seen at the heart and lung clinic per year, and we need to include 3 participants per week, we don't think that we will have a problem to recruit all 238 participants within the study period. However, another pandemic could slow down or interrupt recruitment.

Importance of the study Despite the fact that ARNI have been shown to be beneficial for patients with HFrEF in previous studies, no Africans except a few people living in South Africa were included in these studies. Before implementing ARNI in sub-Saharan Africa, data about efficacy and safety of ARNI in the African population are needed. This interventional pre-post study will deliver this information, encouraging stakeholders and doctors to implement and prescribe this medication in future.

Publication and Dissemination Policy It is intended to publish the results of this study in a peer-reviewed journal in accordance with the journal-specific regulations. Potential conflicts of interest will be listed. Authorship of publications will be based on accepted standards as contained in the guideline "Uniform Requirements for Manuscripts Submitted to Biomedical Journals of the International Committee of Medical Journal Editors" (http://www.icmje.org/urm_main.html). Each person designated as author will have contributed substantially to the intellectual content (conception and design of the study; acquisition, analysis, and interpretation of data) and to the manuscript or the revision including the final approval of the version to be published. In order to disseminate the results, data will be presented at national scientific conferences, and national non-communicable diseases conference. After data analysis, district, regional and national health authorities will receive a letter with all the results. If requested, we will present results personally with health authorities.

Budget justification Total budget is 247'064 SWiss Francs (CHF) 137'236 CHF would be used for salaries, 54240 CHF for consumables, and 22450 CHF for miscellaneous costs. The budget has been approved by the grants offices of the Ifakara Health Institute and Swiss TPH. Funding will be provided by Novartis East Africa.

The costs for guideline directed basic heart failure drugs will be covered by the participants or their health insurance. Sacubitril/valsartan twice a day will be provided by Novartis during the study period (a total of 6'664 tablets Uperio 50mg, 9'996 tablets Uperio 100mg, and 128'520 tablets Uperio 200mg).

ELIGIBILITY:
Inclusion criteria

* Symptomatic heart failure NYHA class II-IV and
* Left ventricular ejection fraction (LVEF) ≤40% and
* Treatment with an ACE Inhibitor or an ARB, beta-blocker, and spironolactone in recommended dosages for at least 3 months, and
* Adherence to this therapy of at least 80%.

Exclusion criteria

* Pregnancy
* Systolic blood pressure of less than 95 mmHg,
* eGFR below 30 ml per minute per 1.73 m2 of body-surface area
* Serum potassium level of more than 5.4 mmol per liter
* History of angioedema
* Unacceptable side effects prior during receipt of ACE inhibitors or ARBs
* Inability to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an improved health status based on a large (≥10 points) or very large (≥20 points) improvement of the Kansas City Cardiomyopathy Questionnaire (KCCQ) summary score (minimum 0, maximum 100) | 10 months
  Higher scores of the Kansas City Cardiomyopathy Questionnaire summary score indicate better outcome

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) summary score (minimum 0, maximum 100) | 5 weeks, 2, 4, 6, and 10 months
  Higher scores of the Kansas City Cardiomyopathy Questionnaire indicate better outcome
New York Heart Association (NYHA) classification (minimum I, maximum IV) | 5 weeks, 2, 4, 6 and 10 months
  Higher classification in the New York Heart Association classification means worse outcome
Distance covered in the 6-minute walking test | 5 weeks, 2, 4, 6 and 10 months
Serum BNP concentration | 10 months
Left ventricular ejection fraction | 6 and 10 months
Proportion of participants with controlled blood pressure | 2 weeks, 5 weeks, and 2, 4, 6, and 10 months
Numbers of hospitalization, death, and loss to follow-up | 10 months

OTHER OUTCOMES:
Number of participants with renal failure, hyperkalemia, angioedema, and hypotension | 10 months
  Number of participants with hyperkalemia, renal failure (defined as a decrease in the estimated glomerular filtration rate (eGFR) of at least 50% or a decrease of at least 30ml per minute per 1.73m2 from time of enrolment to less than 60ml per minute) hypotension (systolic blood pressure <90 mmHg), and angioedema.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel S Mutasingwa, MD, Principal Investigator — Ifakara Health Iistitute
Locations (1):
- Heart and Lung Clinic, St Francis Regional Referral Hospital, Ifakara, Tanzania, Ifakara, Morogoro, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon justified request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12-2027
Access Criteria: IPD will be shared upon justified request

REFERENCES:
- [Background] Senni M, McMurray JJ, Wachter R, McIntyre HF, Reyes A, Majercak I, Andreka P, Shehova-Yankova N, Anand I, Yilmaz MB, Gogia H, Martinez-Selles M, Fischer S, Zilahi Z, Cosmi F, Gelev V, Galve E, Gomez-Doblas JJ, Nociar J, Radomska M, Sokolova B, Volterrani M, Sarkar A, Reimund B, Chen F, Charney A. Initiating sacubitril/valsartan (LCZ696) in heart failure: results of TITRATION, a double-blind, randomized comparison of two uptitration regimens. Eur J Heart Fail. 2016 Sep;18(9):1193-202. doi: 10.1002/ejhf.548. Epub 2016 May 12. PMID 27170530
- [Background] Wang TD, Tan RS, Lee HY, Ihm SH, Rhee MY, Tomlinson B, Pal P, Yang F, Hirschhorn E, Prescott MF, Hinder M, Langenickel TH. Effects of Sacubitril/Valsartan (LCZ696) on Natriuresis, Diuresis, Blood Pressures, and NT-proBNP in Salt-Sensitive Hypertension. Hypertension. 2017 Jan;69(1):32-41. doi: 10.1161/HYPERTENSIONAHA.116.08484. Epub 2016 Nov 14. PMID 27849566
- [Background] Ibrahim NE, Pina IL, Camacho A, Bapat D, Felker GM, Maisel AS, Butler J, Prescott MF, Abbas CA, Solomon SD, Januzzi JL Jr; Prospective Study of Biomarkers, Symptom Improvement and Ventricular Remodeling During Entresto Therapy for Heart Failure (PROVE-HF) Study Investigators. Racial and Ethnic Differences in Biomarkers, Health Status, and Cardiac Remodeling in Patients With Heart Failure With Reduced Ejection Fraction Treated With Sacubitril/Valsartan. Circ Heart Fail. 2020 Nov;13(11):e007829. doi: 10.1161/CIRCHEARTFAILURE.120.007829. Epub 2020 Oct 3. PMID 33016100
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601
- [Background] Thomas M, Khariton Y, Fonarow GC, Arnold SV, Hill L, Nassif ME, Chan PS, Butler J, Thomas L, DeVore AD, Hernandez AF, Albert NM, Patterson JH, Williams FB, Spertus JA. Association between sacubitril/valsartan initiation and real-world health status trajectories over 18 months in heart failure with reduced ejection fraction. ESC Heart Fail. 2021 Aug;8(4):2670-2678. doi: 10.1002/ehf2.13298. Epub 2021 May 1. PMID 33932120
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Raphael DM, Roos L, Myovela V, Mchomvu E, Namamba J, Kilindimo S, Gingo W, Hatz C, Paris DH, Weisser M, Kobza R, Rohacek M. Heart diseases and echocardiography in rural Tanzania: Occurrence, characteristics, and etiologies of underappreciated cardiac pathologies. PLoS One. 2018 Dec 26;13(12):e0208931. doi: 10.1371/journal.pone.0208931. eCollection 2018. PMID 30586432
- [Background] Dokainish H, Teo K, Zhu J, Roy A, AlHabib KF, ElSayed A, Palileo-Villaneuva L, Lopez-Jaramillo P, Karaye K, Yusoff K, Orlandini A, Sliwa K, Mondo C, Lanas F, Prabhakaran D, Badr A, Elmaghawry M, Damasceno A, Tibazarwa K, Belley-Cote E, Balasubramanian K, Islam S, Yacoub MH, Huffman MD, Harkness K, Grinvalds A, McKelvie R, Bangdiwala SI, Yusuf S; INTER-CHF Investigators. Global mortality variations in patients with heart failure: results from the International Congestive Heart Failure (INTER-CHF) prospective cohort study. Lancet Glob Health. 2017 Jul;5(7):e665-e672. doi: 10.1016/S2214-109X(17)30196-1. Epub 2017 May 3. PMID 28476564
- [Background] Chillo P, Mlay J, Akanyirige PW, Majani N, Janabi M, Kaaya S, Hawkins C, Hirschhorn LR. Adapting and usability testing of the Kansas city cardiomyopathy questionnaire (KCCQ) in a heart failure clinic in Tanzania: the Swahili KCCQ. BMC Cardiovasc Disord. 2023 May 6;23(1):242. doi: 10.1186/s12872-023-03265-0. PMID 37149565